CLINICAL TRIAL: NCT02253901
Title: Study of Pharmacokinetic Interaction Between TRUVADA™ and BILR 355 BS Plus Ritonavir
Brief Title: Pharmacokinetic Interaction Between TRUVADA™ and BILR 355 BS Plus Ritonavir in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1188.10
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Ritonavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

ARMS (2):
- TRUVADA with BILR 355 BS and ritonavir (Experimental)
  Interventions: Drug: BILR 355 BS; Drug: Ritonavir; Drug: TRUVADA
- BILR 355 BS in combination with ritonavir (Active Comparator)
  Interventions: Drug: BILR 355 BS; Drug: Ritonavir

INTERVENTIONS:
Drug: BILR 355 BS
Drug: Ritonavir
Drug: TRUVADA
  Arms: TRUVADA with BILR 355 BS and ritonavir

SUMMARY:
Study to determine the pharmacokinetic effect of BILR 355 + ritonavir® on TRUVADA and TRUVADA on BILR 355

ELIGIBILITY:
Inclusion Criteria:

* Males and Females who meet the inclusion/exclusion criteria; females must not be pregnant or nursing, and must agree to use a double-barrier method of birth control (condoms or diaphragm, plus spermicide) throughout the trial (alone or in addition to other methods of birth control such as oral contraceptives)
* Age ≥18 and <60 years
* Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
* Ability to give signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and the local regulations

Exclusion Criteria:

* Current (symptomatic within the last 30 days) and medically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Currently active (symptomatic within the last 30 days) diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within one month prior to administration of study drug or during the trial (review with clinical monitor if questionable)
* Use of drugs within 10 days prior to administration or during the trial, which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation (review with clinical monitor if questionable)
* Participation in another trial with an investigational drug within one month prior to administration or during the trial
* Current smoker
* Alcohol (more than 60 g/day) or drug abuse (positive urine test for illicit prescription or non-prescription drugs or drugs of abuse)
* Recent blood donation (more than 100 mL within 4 weeks prior to administration or during the trial)
* Excessive physical activities (within 1 week prior to study drug administration or during the trial)
* Any laboratory value outside the normal reference range that is of clinical relevance at screening, according to the judgment of the investigator
* Inability to comply with dietary regimen required by the protocol
* Chronic or relevant acute infections
* Infected with hepatitis B or hepatitis C viruses (defined as either being hepatitis B surface antigen, or hepatitis C antibody positive)
* HIV-1 infected as defined by a positive HIV ELISA test

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2005-03; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from 0 to 24 hours at steady state of the analyte in plasma (AUC0-24h,ss) | up to 24 h after treatment

SECONDARY OUTCOMES:
Apparent clearance of the analyte in plasma following extravascular administration at steady state (CL/F,ss) | up to day 18 after start of treatment
Time from dosing to the maximum concentration of the analyte in plasma at steady state (tmax,ss) | up to day 18 after start of treatment
Measured concentration of the analyte in plasma 24 hours post last dose at steady state (Cp24h, ss) | up to 24 h after treatment
Terminal half-life of of the analyte in plasma in the plasma at steady state (t1/2, ss) | up to day 18 after start of treatment
Apparent volume of distribution of of the analyte in plasma during the terminal phase λz at steady state following an extravascular dose (Vz/F,ss) | up to day 18 after start of treatment
Area under the concentration-time curve from 0 to 24 hours of ritonavir in plasma (AUC0-24h) | up to 24 h after treatment
Maximum measured concentration of ritonavir in plasma (Cmax) | up to 24 h after treatment
Number of subjects with clinically relevant changes in clinical laboratory tests | up to day 28 after start of treatment
Number of subjects with clinically relevant changes in vital signs (blood pressure, pulse rate) | up to day 28 after start of treatment
Number of subjects with adverse events | Up to 7 weeks